CLINICAL TRIAL: NCT02002572
Title: Quantification, Analysis and Simulation of Facial Mimics Movements
Acronym: SIMOVI-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Regional Council Picardie, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI11-DR-DAKPE; 2011-A00532-39 (Other: ID-RCB)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mimic Facial Muscles
Keywords: Facial Mimic Muscle; MRI; Segmentation; Three dimensional assessment; Motion capture; Movement analysis; Digital Image Correlation
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Motion Capture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mimic facial muscle from 3T MRI data (Experimental)
  Interventions: Other: Magnetic Resonance Imaging (MRI), Surface scan, Motion capture, Digital Image Correlation

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI), Surface scan, Motion capture, Digital Image Correlation

SUMMARY:
The SIMOVI project is a collaboration between our Department of Maxillofacial Surgery (CHU Amiens) and the Biomechanical bioengineer Research Department and Roberval Labs (Technological University of Compiègne). The question raised is the extent to which a facial mimic can be evaluated objectively. In today's clinical practice, the investigators use grading systems based on muscular scale or testing, in order to evaluate a facial muscular disorder. This assessment remains subjective because the investigators are deducing from surfacing cutaneous deformations the movement quality of the solicited muscle.

This qualitative approach is therefore an approximate approach and deserves to be better thought to plan a surgical treatment which involves mimic facial muscle (as rehabilitation of facial palsy, cleft palate for example), to monitor the results, and to follow the recovery and progress in physiotherapy care.

The aim of this study is to correlate external soft tissue movement (essentially cutaneous) during facial mimic with internal movement (essentially facial mimic muscle) using qualitative and QUANTITATIVE indicators, and to perform a biomechanical model of selected mimic face's movement using the precedent data.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subject
* Ability to provide informed consent

Exclusion Criteria:

* Facial pathology
* Facial trauma
* Pregnant or breastfeeding.
* Contraindications to MRI

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08-08 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Morphometric assessment of mimic facial muscle from 3T MRI data | 30 min
  The aim is to valid a method to identify, describe and measure the mimic facial muscles in 3 Tesla MRI. Through particular MRI acquisition developed especially for mimic facial muscle from routine acquisition, Morphometrics properties are calculated as length, volume, thickness and cross physiological section area.

SECONDARY OUTCOMES:
Three dimensional quantitative analysis of mimics through motion capture | 01 hour
  A VICON motion capture system with the Nexus 1.7.1 software will be used to capture expressive facial movements at a 120 Hz sample rate with 7 T160 cameras and 2 MX30 cameras. Markers of a diameter of 1.5 mm will be placed on the face. The localization of the markers is related to the muscles involved in the movements we want to study.
  After data capture, we build and reconstruct our model. We chose a neutral pose as reference. The best parameters for the reconstruction will be determined. Kinematic parameters will be the markers displacement.
Three dimensional quantitative mimic facial analysis with surface scan. | 01 hour
  Three-dimensional image captured with a MH WHALE 3D Scanner.
Three dimensional analysis with Digital Image Correlation | 01 hour
  Recording three-dimensional images of the deformations of the face by two pairs of Pike CCD cameras from Allied Vision Technologies, with Schneider Xenoplan 2.0/28mm Lens, positioned on both sides of the face.
  The calibration and the image processing will be made with the software suite VIC-SNAP, VIC-3D and 3D Fusion (Correlated Solutions)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, MD, phD, Study Director — Department of Maxillofacial Surgery, Amiens University Hospital; Stéphanie DAKPE, MD, Principal Investigator — Department of Maxillofacial Surgery, Amiens University Hospital
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

REFERENCES:
- [Background] Autuori B, Bruyere-Garnier K, Morestin F, Brunet M, Verriest JP. Finite element modeling of the head skeleton with a new local quantitative assessment approach. IEEE Trans Biomed Eng. 2006 Jul;53(7):1225-32. doi: 10.1109/TBME.2006.872812. PMID 16830926
- [Background] Barbarino GG, Jabareen M, Trzewik J, Nkengne A, Stamatas G, Mazza E. Development and validation of a three-dimensional finite element model of the face. J Biomech Eng. 2009 Apr;131(4):041006. doi: 10.1115/1.3049857. PMID 19275435
- [Background] Bensamoun SF, Ringleb SI, Littrell L, Chen Q, Brennan M, Ehman RL, An KN. Determination of thigh muscle stiffness using magnetic resonance elastography. J Magn Reson Imaging. 2006 Feb;23(2):242-7. doi: 10.1002/jmri.20487. PMID 16374878
- [Background] Bensamoun S, Stevens L, Fleury MJ, Bellon G, Goubel F, Ho Ba Tho MC. Macroscopic-microscopic characterization of the passive mechanical properties in rat soleus muscle. J Biomech. 2006;39(3):568-78. doi: 10.1016/j.jbiomech.2004.04.036. PMID 16389097
- [Background] Brix M, Raphael B. [Labial function]. Ann Chir Plast Esthet. 2002 Oct;47(5):357-69. doi: 10.1016/s0294-1260(02)00129-2. French. PMID 12449863
- [Background] Burres SA. Facial biomechanics: the standards of normal. Laryngoscope. 1985 Jun;95(6):708-14. doi: 10.1288/00005537-198506000-00013. PMID 3999905
- [Background] Burres SA. Objective grading of facial paralysis. Ann Otol Rhinol Laryngol. 1986 May-Jun;95(3 Pt 1):238-41. doi: 10.1177/000348948609500306. PMID 3717849
- [Background] Burres S, Fisch U. The comparison of facial grading systems. Arch Otolaryngol Head Neck Surg. 1986 Jul;112(7):755-8. doi: 10.1001/archotol.1986.03780070067015. PMID 3707739
- [Background] Cacou C, Greenfield BE, Hunt NP, McGrouther DA. Patterns of coordinated lower facial muscle function and their importance in facial reanimation. Br J Plast Surg. 1996 Jul;49(5):274-80. doi: 10.1016/s0007-1226(96)90155-1. PMID 8774240
- [Background] Chabanas M, Payan Y, Marecaux C, Swider P, Boutault F Comparison of linear and non linear soft tissue models with post-operative CT scan in maxillofacial surgery Lecture notes in computer science 2004, vol 3078, 19-27
- [Background] Chevallier AM.Rééducation des paralysies faciales centrales et périphériques Encyclopédie Médico-Chirurgicale, Paris Kinésithérapie 26463 B10 5-1990, 16 p
- [Background] Coulson SE, Croxson GR, Gilleard WL. Three-dimensional quantification of
- [Background] Croxson G, May M, Mester SJ. Grading facial nerve function: House-Brackmann versus Burres-Fisch methods. Am J Otol. 1990 Jul;11(4):240-6. PMID 2399941
- [Background] Duchenne de Boulogne.La mécanique des passions. Paris ,1855
- [Background] Ekman P, Friesen W.V .Unmasking the face: A guide to recognizing emotions from facial clues Consulting psychologists press (Palo Alto, Californie 1984)
- [Background] Ermiane.R.Jeux musculaires et expressions du visage.Paris : Le François
- [Background] Farrugia ME, Bydder GM, Francis JM, Robson MD. Magnetic resonance imaging of facial muscles. Clin Radiol. 2007 Nov;62(11):1078-86. doi: 10.1016/j.crad.2007.05.003. Epub 2007 Aug 9. PMID 17920867
- [Background] Gladilin E, Zackav S, Deufhard P, HEGE HC.Towards a realistic simulation of individual facial mimics Stuttgart, Germany, November 21-23, 2001
- [Background] Ho Ba Tho MC Bone and joints modelling with individualised geometric and mechanical properties derived from medical images. Computer Mechanics and Engineering Sciences (2003) 4: 3&4. 489-496
- [Background] Hontanilla B, Auba C. Automatic three-dimensional quantitative analysis for evaluation of facial movement. J Plast Reconstr Aesthet Surg. 2008;61(1):18-30. doi: 10.1016/j.bjps.2007.03.037. Epub 2007 Jun 13. PMID 17569607
- [Background] House JW, Brackmann DE. Facial nerve grading system. Otolaryngol Head Neck Surg. 1985 Apr;93(2):146-7. doi: 10.1177/019459988509300202. No abstract available. PMID 3921901
- [Background] Isono M, Murata K, Tanaka H, Kawamoto M, Azuma H. An objective evaluation method for facial mimic motion. Otolaryngol Head Neck Surg. 1996 Jan;114(1):27-31. doi: 10.1016/S0194-59989670279-6. PMID 8570246
- [Background] Deng J, Newton NM, Hall-Craggs MA, Shirley RA, Linney AD, Lees WR, Rodeck CH, McGrouther DA. Novel technique for three-dimensional visualisation and quantification of deformable, moving soft-tissue body parts. Lancet. 2000 Jul 8;356(9224):127-31. doi: 10.1016/S0140-6736(00)02449-1. PMID 10963249
- [Background] Kleinheinz J, Joos U. Imaging of cartilage and mimic muscles with MRI: anatomic study in healthy volunteers and patients with unilateral cleft lip and palate. Cleft Palate Craniofac J. 2001 Jul;38(4):291-8. doi: 10.1597/1545-1569_2001_038_0291_iocamm_2.0.co_2. PMID 11420008
- [Background] Lacide.M, Chevallier .AM Evaluation clinique de la fonction musculaire.
- [Background] Le Double AF.Traité des variations du système musculaire de l'homme1897, Paris : Schleicher frères
- [Background] Linstrom CJ, Silverman CA, Susman WM. Facial-motion analysis with a video and computer system: a preliminary report. Am J Otol. 2000 Jan;21(1):123-9. doi: 10.1016/s0196-0709(00)80086-1. PMID 10651446
- [Background] Luboz V, Chabanas M, Swider P, Payan Y. Orbital and maxillofacial computer aided surgery: patient-specific finite element models to predict surgical outcomes. Comput Methods Biomech Biomed Engin. 2005 Aug;8(4):259-65. doi: 10.1080/10255840500289921. PMID 16298848
- [Background] Meier-Gallati V, Scriba H, Fisch U. Objective scaling of facial nerve function based on area analysis (OSCAR). Otolaryngol Head Neck Surg. 1998 Apr;118(4):545-50. doi: 10.1177/019459989811800419. PMID 9560110
- [Background] Paletz JL, Manktelow RT, Chaban R. The shape of a normal smile: implications for facial paralysis reconstruction. Plast Reconstr Surg. 1994 Apr;93(4):784-9; discussion 790-1. PMID 8134437
- [Background] Payan Y, Chabanas M, Pelorson X, Vilain C, Levy P, Luboz V, Perrier P. Biomechanical models to simulate consequences of maxillofacial surgery. C R Biol. 2002 Apr;325(4):407-17. doi: 10.1016/s1631-0691(02)01443-9. English, French. PMID 12161921
- [Background] Pessa JE, Zadoo VP, Adrian EK Jr, Yuan CH, Aydelotte J, Garza JR. Variability of the midfacial muscles: analysis of 50 hemifacial cadaver dissections. Plast Reconstr Surg. 1998 Nov;102(6):1888-93. doi: 10.1097/00006534-199811000-00013. PMID 9810983
- [Background] Poirrier P, Charpy A.Traité d'anatomie humaine..Myologie, vol. 2, 1901, Paris, Masson
- [Background] Rouvière H .Anatomie humaine descriptive, topographique et fonctionnelle.Tome 1, Tête et cou, 15e édition
- [Background] Rubin LR. The anatomy of a smile: its importance in the treatment of facial paralysis. Plast Reconstr Surg. 1974 Apr;53(4):384-7. doi: 10.1097/00006534-197404000-00002. No abstract available. PMID 4815693
- [Background] Sangeux M, Marin F, Charleux F, Durselen L, Ho Ba Tho MC. Quantification of the 3D relative movement of external marker sets vs. bones based on magnetic resonance imaging. Clin Biomech (Bristol). 2006 Nov;21(9):984-91. doi: 10.1016/j.clinbiomech.2006.05.006. Epub 2006 Jul 17. PMID 16844273
- [Background] Sobotta.Atlas d'anatomie humaine - Tome 13 - Edition française.Edition Médicale Internationale, 1994
- [Background] Testud L.Traité d'anatomie humaine.1899, Paris
- [Background] Tomat LR, Manktelow RT. Evaluation of a new measurement tool for facial paralysis reconstruction. Plast Reconstr Surg. 2005 Mar;115(3):696-704. doi: 10.1097/01.prs.0000152431.55774.7e. PMID 15731666
- [Background] Tran HV, Charleux F, Rachik M, Ehrlacher A, Ho Ba Tho MC. In vivo characterization of the mechanical properties of human skin derived from MRI and indentation techniques. Comput Methods Biomech Biomed Engin. 2007 Dec;10(6):401-7. doi: 10.1080/10255840701550287. Epub 2007 Sep 24. PMID 17891674
- [Background] Tran H V (2007) Determination of the mechanical properties of the skin in vivo. PhD Dissertation, Université de Technologie de Compiègne
- [Background] Wang S, Yang J. Simulating cranio-maxillofacial surgery based on mixed-element biomechanical modelling. Comput Methods Biomech Biomed Engin. 2010 Jun;13(3):419-29. doi: 10.1080/10255840903317386. PMID 20077239
- [Background] Wang S, Yang J, Gee JC. Advances in collision detection and non-linear finite mixed element modelling for improved soft tissue simulation in craniomaxillofacial surgical planning. Int J Med Robot. 2010 Mar;6(1):28-41. doi: 10.1002/rcs.286. PMID 19946886
- [Background] Wood DA, Hughes GB, Secic M, Good TL. Objective measurement of normal facial movement with video microscaling. Am J Otol. 1994 Jan;15(1):61-5. PMID 8109633
- [Background] Hartl DM, Kolb F, Bretagne E, Bidault F, Sigal R. Cine-MRI swallowing evaluation after tongue reconstruction. Eur J Radiol. 2010 Jan;73(1):108-13. doi: 10.1016/j.ejrad.2008.10.005. Epub 2008 Dec 16. PMID 19091505
- [Background] Farrugia ME, Robson MD, Clover L, Anslow P, Newsom-Davis J, Kennett R, Hilton-Jones D, Matthews PM, Vincent A. MRI and clinical studies of facial and bulbar muscle involvement in MuSK antibody-associated myasthenia gravis. Brain. 2006 Jun;129(Pt 6):1481-92. doi: 10.1093/brain/awl095. Epub 2006 May 3. PMID 16672291
- [Result] https://doi.org/10.1080/10255842.2014.931142
- [Result] Sarhan FR, Olivetto M, Ben Mansour K, Neiva C, Colin E, Choteau B, Marie JP, Testelin S, Marin F, Dakpe S. Quantified analysis of facial movement: A reference for clinical applications. Clin Anat. 2023 Apr;36(3):492-502. doi: 10.1002/ca.23999. Epub 2023 Jan 24. PMID 36625484